CLINICAL TRIAL: NCT06093542
Title: A Randomised, Single-blind, Single Center, Placebo-controlled, Phase I Study to Assess the Safety, Tolerability, and Pharmacokinetics of AZD7503 Following Multiple Subcutaneous Dose Administration in Healthy Japanese Participants.
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of AZD7503 in Japanese Healthy Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D9230C00005
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Heathy Participants
Keywords: Non-alcoholic Fatty Liver Disease cirrhosis; N-acetyl galactosamine-conjugated antisense oligonucleotide; HSD17B13 protein

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The study is single blind where the study site staff including the investigator will remain blinded during the clinical conduct of a given cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD7503 (Experimental): Participants will subcutaneously receive AZD7503.
  Interventions: Drug: AZD7053
- Placebo (Placebo Comparator): Participants will subcutaneously receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD7053 — Randomised participants will receive AZD7503 subcutaneously.
  Arms: AZD7503
Drug: Placebo — Randomised participants will receive placebo subcutaneously.
  Arms: Placebo

SUMMARY:
The study will evaluate the safety, tolerability, and the pharmacokinetics (PK) of AZD7503 following multiple subcutaneous doses in healthy Japanese participants.

DETAILED DESCRIPTION:
This is a Phase I, randomised, single-blind, placebo-controlled study. The healthy Japanese participants will receive randomly (3:1) either AZD7503 or placebo subcutaneously.

The study will comprise of:

* A screening period of 28 days.
* Randomization on Day 1.
* A 9-week Treatment Period. Dose 1 will be administered on Day 1. Dose 2 will be administered at the study site on Day 29. Dose 3 will be administered on Day 57.
* A follow-up period of 10 week after last dose of study intervention.
* The total duration of the study will be 23 weeks

ELIGIBILITY:
Inclusion Criteria:

* For Japanese participants: A Japanese participant is defined as having both parents and 4 Japanese grandparents as confirmed by the interview. This includes second and third generation Japanese whose parents or grandparents are living in a country other than Japan. Participants must have suitable veins for cannulation.
* Females must be of non-childbearing potential.
* Males and females must adhere to the contraception methods.
* Have a Body mass index between 18 and 30 kg/m2 inclusive.

Exclusion Criteria:

* History of any clinically significant disease or disorder in the investigator's opinion.
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure or trauma.
* Any abnormal laboratory values, clinical chemistry, hematology or urinalysis results, vital signs, Electrocardiography.
* Any clinically significant cardiovascular event.
* Participants with known autoimmune disease or on-treatment with immune-modulatory drugs.
* Any positive result at the Screening Visit for serum Hepatitis B surface antigen, hepatitis C antibody and Human Immunodeficiency virus.
* Confirmed COVID-19 infection during screening as per local guidelines.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity.
* Use of any prescribed or nonprescribed medication.
* History of major bleed or high-risk of bleeding diathesis.
* Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of study intervention.
* Participants who have previously received AZD7503 or any investigational drug targeting HSD17B13.
* Vulnerable participants.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | From Screening (Day -28) until Follow-up Day 127 (10 weeks post last dose)
  The safety and tolerability after multiple doses of AZD7503 in healthy Japanese participants will be evaluated.

SECONDARY OUTCOMES:
Maximum plasma drug concentration (Cmax) | Day 1, Day 2, Day 3, Day 5, Day 15, Day 29, Day 57, Day 58, and Day 59
  The Cmax after administration of multiple doses of AZD7503 in healthy Japanese participants will be evaluated.
Are under plasma concentration-time curve from time 0 to the last quantifiable concentration (AUClast) | Day 1, Day 2, Day 3, Day 5, Day 15, Day 29, Day 57, Day 58, and Day 59
  The AUClast after administration of multiple doses of AZD7503 in healthy Japanese participants will be evaluated.
Area under plasma concentration-time curve from time 0 to infinity (AUCinf) | Day 1, Day 2, Day 3, Day 5, Day 15, Day 29, Day 57, Day 58, and Day 59
  The AUCinf after administration of multiple doses of AZD7503 in healthy Japanese participants will be evaluated.
Area under plasma concentration-time curve during a dosing interval (AUCtau) | Day 1, Day 2, Day 3, Day 5, Day 15, Day 29, Day 57, Day 58, and Day 59
  The AUCtau after administration of multiple doses of AZD7503 in healthy Japanese participants will be evaluated.
Amount of analyte excreted into the urine (Ae) | Day 1, Day 2, Day 3, Day 58, and Day 59
  The Ae after administration of multiple doses of AZD7503 in healthy Japanese participants will be evaluated.
Fraction of the dose excreted unchanged in urine (Fe) | Day 1, Day 2, Day 3, Day 58, and Day 59
  The Fe after administration of multiple doses of AZD7503 in healthy Japanese participants will be evaluated.
Plasma concentration of AZD7503 | Day 1, Day 2, Day 3, Day 58, and Day 59
  The plasma concentration after administration of multiple doses of AZD7503 in healthy Japanese participants will be evaluated.
Plasma concentration of unconjugated antisense oligonucleotide (ASO) | Day 1, Day 2, Day 3, Day 58, and Day 59
  The plasma concentration of unconjugated ASO at specified timepoints after administration of multiple doses of AZD7503 in healthy Japanese participants will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Sumida-ku, Japan

REFERENCES:
- See also: Redacted_CSR Synopsis_D9230C00005 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9230C00005&attachmentIdentifier=54bc5a37-9983-4626-99ba-9b0dbcb0705d&fileName=Redacted_CSR_Synopsis_D9230C00005.pdf&versionIdentifier=